CLINICAL TRIAL: NCT06316986
Title: Performance of the NGPOD® Device in Verifying the Correct Position in the Stomach of the Naso- or Oro- Gastric Tube in Intensive Care : Prospective Monocentric Clinical Investigation
Brief Title: Performance of the NGPOD® Device in Verifying the Correct Position in the Stomach of the Naso- or Oro- Gastric Tube in Intensive Care.
Acronym: NGPOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2023-A02294-41
Record Dates: First submitted 2024-01-12; First posted 2024-03-19 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Intensive Care; Nutrition
Keywords: naso gastric tube; oro gastric tube; PH

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients requiring an orogastric or nasogastric tube (Experimental)
  Interventions: Diagnostic Test: pH indication with NGPOD

INTERVENTIONS:
Diagnostic Test: pH indication with NGPOD — The NGPOD sensor is inserted into the naso- or oro-gastric tube, then reconnected to the NGPOD handheld device, and the pH measurement is taken within 15 seconds.
  When the 15 seconds have elapsed, the pH button is pressed. If the green LED lights up and the pH indicates a value < 5.5, the sensor tip is in a pH environment associated with the stomach.
  If the red LED lights up, the sensor tip is in a pH environment NOT associated with the stomach.

SUMMARY:
In the Intensive Care Unit (ICU), scientific societies recommend starting enteral nutrition within 48 hours of admission, if oral nutrition is not available, in order to limit undernutrition. In patients who are sedated, have swallowing problems or cannot ensure adequate caloric intake, it is essential to insert a feeding tube, usually a nasogastric or orogastric tube for the first few weeks.

Placement of a naso- or oro-gastric tube in the intensive care unit is a frequent procedure, and considered to be straightforward. It is usually performed blindly, at the patient's bedside, by a nurse or doctor, according to a departmental protocol or the recommendations of learned societies.

Nevertheless, a number of complications have been reported with naso- or oro-gastric tubes, linked in particular to a route outside the digestive tract : malpositioning/coiling of the tube, epistaxis, sinusitis. The most frequent and potentially severe complications are malpositions in the tracheobronchial tree.

Radiographic control is currently considered in France and by certain learned societies to be the reference method for verifying correct positioning of the probe in the stomach (at the prepyloric antral level). However, thoracic radiography has a number of drawbacks : In intensive care risk of accidental displacement of other medical devices,irradiation, difficulty of interpretation, delay in obtaining the image, time-consuming work for qualified personnel.

An alternative technique using the NGPOD device is proposed as a method of checking the correct positioning of the probe in the stomach. This system enables immediate, rapid (15 seconds), simple and automatic testing at the patient's bedside. The device provides a visual indication of the pH detected at the tip of the gastric tube. The test result is given in binary form: Yes (green signal, probe in stomach) / No (red signal, probe incorrectly positioned).

Study hypothesis and prospects: To make an initial estimate of the sensitivity and specificity of the NGPOD system for checking the positioning of the naso- or oro-gastric tube in the stomach, compared with the recognized gold standard, the chest X-ray.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in intensive care
* Patients aged 18 or over with no upper age limit
* Patients admitted to intensive care with a nasogastric or orogastric tube placed in the operating room (not controlled by radiography) or for whom the placement of a gastric tube in intensive care is indicated.
* Consent to research participation

Exclusion Criteria:

* Patients undergoing limitation and discontinuation of active therapies
* Patients with contraindications to blind gastric tube placement (recent esophageal or gastric surgery, ENT lesions, uncontrolled upper GI bleeding, esophageal or gastric cancer)
* Patients under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Ability of the NGPOD device to detect correct positioning of the gastric tube. | Up to one Day
  Comparison of NGPOD and chest X-ray results.

SECONDARY OUTCOMES:
Probe malpositioning | Up to one Day
  collection of malpositioning site
Time to validate correct positioning of gastric tube | Up to one Day
  This time will be calculated as the difference between the following times:
  * T0: time when the SNG is installed and checked by auscultation.
  * TNGPOD: time when SNG positioning is estimated by the NGPOD system.
  * TRT: time when the positioning of the SNG is estimated in place in the stomach on the chest X-ray, by a doctor.
  * TRTDEF: time when the positioning of the SNG is estimated in place by the doctor on the 2nd x-ray, in the event that the probe is not visualized on the 1st x-ray. In the event that the X-ray does not allow the gastric tube to be visualized, the technical parameters of the X-ray and/or opacification of the tube will be modified, and a new X-ray will be taken and interpreted.
Evaluation of the "simplicity" of the procedures for using and interpreting the NGPOD system | Up to one Day
  Scale from 0 to 10- 0 for easy and 10 for very difficult
x-ray manipulators time | "through study completion, an average of 1 year"
  Evaluation of the working time of radiology manipulators
Adverse events occurring during the study period | "through study completion, an average of 1 year"
Ability of the NGPOD device to detect correct gastric tube positioning in a subgroup of patients | Up to one Day
  * patients treated with proton pump inhibitors
  * patients who received nutrition within 6 hours prior to tube insertion

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Marie Lannelongue, Le Plessis-Robinson, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Singer P, Blaser AR, Berger MM, Alhazzani W, Calder PC, Casaer MP, Hiesmayr M, Mayer K, Montejo JC, Pichard C, Preiser JC, van Zanten ARH, Oczkowski S, Szczeklik W, Bischoff SC. ESPEN guideline on clinical nutrition in the intensive care unit. Clin Nutr. 2019 Feb;38(1):48-79. doi: 10.1016/j.clnu.2018.08.037. Epub 2018 Sep 29. PMID 30348463
- [Background] Metheny NA, Meert KL, Clouse RE. Complications related to feeding tube placement. Curr Opin Gastroenterol. 2007 Mar;23(2):178-82. doi: 10.1097/MOG.0b013e3280287a0f. PMID 17268247
- [Background] Metheny NA, Krieger MM, Healey F, Meert KL. A review of guidelines to distinguish between gastric and pulmonary placement of nasogastric tubes. Heart Lung. 2019 May-Jun;48(3):226-235. doi: 10.1016/j.hrtlng.2019.01.003. Epub 2019 Jan 18. PMID 30665700